CLINICAL TRIAL: NCT02969850
Title: A New Paradigm for Vitamin D Sufficiency: A 6-month, Randomized, Double-blind, Placebo-controlled Study to Investigate Vitamin D Status in Elderly Caucasian Women
Brief Title: A New Paradigm for Vitamin D Sufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 19-00873
Record Dates: First submitted 2016-11-10; First posted 2016-11-21 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: New Biomarkers for Measuring Vitamin D Level
Keywords: vitamin D supplementation; calcium supplementation
MeSH Terms: interventions — Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D Supplementation (Experimental): Participant will receive initial dose of 2400, 3600, or 4800 IU of vitamin D3, based on her serum vitamin D level. Dose will be adjusted at 3 month visit to maintain serum vitamin D level at a desirable level. If subject has insufficient dietary calcium intake, calcium supplementation will be provided in the form of one 600mg CaCO3 pill to achieve a total calcium intake of 1200mg/day.
  Interventions: Dietary Supplement: Vitamin D Supplementation; Dietary Supplement: Calcium
- Placebo (Placebo Comparator): Participant will receive a placebo. If subject has insufficient dietary calcium intake, calcium supplementation will be provided in the form of one 600mg CaCO3 pill to achieve a total calcium intake of 1200mg/day.
  Interventions: Other: Placebo; Dietary Supplement: Calcium

INTERVENTIONS:
Dietary Supplement: Vitamin D Supplementation — Subjects in this group will receive initial dose of 2400, 3600, or 4800 IU of vitamin D3, based on her serum vitamin D level. Dose will be adjusted at 3 month visit to maintain serum vitamin D level at a desirable level.
  Arms: Vitamin D Supplementation
Other: Placebo — Subjects in this group will receive a placebo.
  Arms: Placebo
Dietary Supplement: Calcium — If dietary calcium intake is insufficient in participants of either group, they will be given a calcium supplement in the form of one 600mg pill of CaCO3 to bring them up to an intake of 1200mg/day.

SUMMARY:
Although the African-American (AA) population tends to have lower serum 25(OH)D levels compared to whites, there is no evidence that the lower 25(OH)D levels in African-Americans are harmful. In fact, skeletal health is superior in AA. It is clear that total serum 25(OH)D concentrations do not reflect the same risk/benefit ratio in AA compared to white women and is, therefore, an inappropriate biomarker in this population.

The investigators wish to investigate whether free 25(OD)D and Vitamin D Metabolite Ratio (VMR, ratio of 25(OH)D to 24,25(OH)2D) are preferable biomarkers to total 25(OH)D. The investigators propose a six month randomized double blinded study.

DETAILED DESCRIPTION:
The specific aims of this study are as follows:

1. To establish that free 25(OH)D and VMR are similar in black and white populations.
2. To characterize the relationships between free 25(OH)D and VMR and two measures of bone health (PTH and BMD) in black and white women.
3. To evaluate whether the relationship of free 25(OH)D (and in parallel analyses, VMR) and bone health are stronger than those based on total 25(OH)D.
4. To evaluate whether free 25(OH)D and VMR respond to vitamin D intake (dose-response) in a similar manner to total 25(OH)D.

The study population is postmenopausal Caucasian women age 60 and older. This six month study includes four visits. These results will be compared to those from a study in AA women which the investigators are also completing.

There are two study groups. One group will receive vitamin D supplementation, the other a placebo. Subjects will be asked to refrain from taking outside Vitamin D supplements for the duration of the study. If the subject is eligible based on the results from the first two visits, the subject will be randomized into one of these two groups. Randomized subjects will be taking the vitamin D or placebo for a period of 6 months and will have one visit at the 3 month mark and a final visit at the 6 month mark.

At the 3-month visit, the following procedures will be conducted: obtain interim medical and travel history, vital signs, weight, and height measured by the Harpenden Stadiometer, record adverse events and concomitant medications, Fasting blood collection: total 25(OH)D (by Diasorin), PTH, serum calcium and creatinine, Fasting urine collection for calcium and creatinine, and questionnaires: calcium food frequency questionnaire, quality of life questionnaire, falls and flu questionnaires. Subjects will be instructed on how to collect a 24-hour urine sample (for final visit) and collection container will be dispensed. Unused study supplements will be collected and counted, and study supplements will be dispensed based on serum 25(OH)D level algorithm.

At the 6-month visit, in addition to what is completed at the 3-month visit, the following procedures will also be conducted:24-hour urine calcium, sodium, oxalate and creatinine; mini-mental health examination; physical performance examination (SPPB); and a physical activity questionnaire. Unused study supplements will be collected and counted. No further supplementation will be provided.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory women older than 60 years of age. Women who are ambulatory with an assistive device such as cane or walker may be included. LMP must be > 5 years ago.
2. Self declared as white.
3. 20 nmol/L < Serum 25(OH)D level < 65 nmol/L.
4. Willingness to take study drug and participate for 6 months in the trial.
5. Willingness to refrain from the use of self-administered Vitamin D and Calcium supplements during the trial.

Exclusion Criteria:

1. Serum 25(OH)D levels ≤ 20 nmol/L or ≥ 65 nmol/L.
2. BMD total hip below -2.5 standard deviation (using NHANES III adult young white men and women as the point of reference) or history of osteoporotic fracture.
3. Moderate to severe fracture in one or more vertebrae by Instant Vertebral Assessment on DXA.
4. Treatment with HRT, SERMs, calcitonin, PTH, strontium ranelate, androgens, bisphosphonates, Denosumab or anabolic steroids during 6 months prior to entry.
5. Use of systemic corticosteroids (oral or IV) within the last year at an average dose of greater than 5 mg per day of oral prednisone or equivalent for a period of three months or more prior to screening.
6. Mini-Mental State Exam score below 21
7. Hypercalcemia (serum calcium > 10.6 mg/dl) or history of primary hyperparathyroidism.
8. History of hypercalciuria, kidney stones, or 24hr urine calcium >261 mg/day on screening.
9. History of chronic liver disease, chronic renal insufficiency (GFR<30), Parkinson's, metabolic bone disease (Hyperparathyroidism, Hypoparathyroidism, Paget's disease, Fibrous osteodystrophy, Rickets, Osteomalacia, Osteosclerosis), hematologic tumors, rheumatologic disease requiring steroids, conditions that influence vitamin D absorption like celiac disease and irritable bowel disease, malabsorption or new diagnosis or active treatment of cancer 12 months prior to inclusion.
10. Use of medications that influence bone metabolism (e.g. anticonvulsants).
11. Significant deviation from normal in either: history, physical examination or laboratory tests as evaluated by the Principle Investigator. Participants with a history of uncontrolled hypertension, uncontrolled diabetes, hypercalciuria, nephrolithiasis and active sarcoidosis or tuberculosis will also be excluded.
12. Participation in another investigational trial 30 days prior to screening.
13. Spinal disease that affects interpretation of bone densitometry like scoliosis with a Cobb angle greater than 15o, history of surgery at lumbosacral spine.
14. Bilateral hip replacement.
15. Currently smoking more than 10 cigarettes daily.
16. Currently consuming more than 2 units of alcohol daily. (One unit is equivalent to a standard glass of beer (285ml), a single measure of spirits (30ml), a medium-sized glass of wine (120ml), or 1 measure of an aperitif (60ml)
17. Unable to perform DXA due to excessive body girth/width. Body width on DXA > 25 cm.
18. Patients who are deemed unsafe to perform muscular function testing as evaluated by the investigator.
19. Class III obesity.

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Compare free 25(OH)D levels in Caucasian women (current study) and AA women (from prior study) | baseline
  VDBP will be measured and free 25(OH)D calculated
Compare Vitamin D metabolite ratio (VMR) in Caucasian women (current study) and AA women (from prior study) | baseline
  serum 24,25(OH)2D and serum 25(OH)D will be measured and VMR calculated

SECONDARY OUTCOMES:
Relationship between free 25(OH)D and two measures of bone health (PTH and BMD) | baseline
  Relationships will be assessed via correlation and regression analyses
Relationship between VMR and two measures of bone health (PTH and BMD) | baseline
  Relationships will be assessed via correlation and regression analyses
Relationship between vitamin D intake and Change in Physical Performance Assessment (SPPB) | baseline and 6 months
  Relationships will be assessed via Mixed-Effects Model for Repeated Measures (MMRM)

CONTACTS AND LOCATIONS:
Overall Officials: John Aloia, MD, Principal Investigator — Winthrop University Hospital; Mageda Mikhail, MD, Study Director — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: No